CLINICAL TRIAL: NCT05652920
Title: A Phase Ib/II, Open-Label, Multi-Center Study to Investigate the Safety, PK, and Efficacy of Ori-C101 in Advanced Hepatocellular Carcinoma (HCC) Patients (BEACON)
Brief Title: Ori-C101Chimeric Antigen Receptor (CAR) Modified T Cells for the Treatment of HCC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OriCell Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ori-C101-P1
Record Dates: First submitted 2022-11-27; First posted 2022-12-15 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ori-C101 ( GPC3-directed chimeric antigen receptor modified T cells ) (Experimental)
  Interventions: Biological: Ori-C101

INTERVENTIONS:
Biological: Ori-C101 — Hepatic arterial infusion

SUMMARY:
This is a Phase I, open-label, multi-center study to assess the safety, pharmacokinetics, and preliminary efficacy of GPC3-directed chimeric antigen receptor modified T cells injection (Ori-C101) in Advanced Hepatocellular Carcinoma(HCC).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed pathologic or radiologic diagnosis of HCC ;
2. Tumor tissue GPC3 expression positive by immunohistochemistry(IHC) at the local laboratory (Tumor samples ≤1 years prior to ICF signature are acceptable), if no archived tumor tissue samples, tumor biopsy is required for GPC3 expression test;
3. Unresectable stage B (intermediate) or C (advanced) HCC according to the Barcelona Clinic Liver Cancer (BCLC) staging. If stage B, must have progressed after, or not be eligible for, surgical or locoregional therapy;
4. Received at least two prior line of systemic therapy (included but not limited to target therapy, immunotherapy or chemotherapy) with radiologic disease progression during or following systemic therapy;
5. Child-Pugh A or B7, no history of hepatic encephalopathy;
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 at the time of ICF signature;
7. Estimated life expectancy of minimum of 12 weeks;
8. Must have at least 1 target lesion

Exclusion Criteria:

1. Central nervous system metastatic disease, leptomeningeal disease, or metastatic cord compression;
2. Prior bone marrow or organ transplantation;
3. Have a history of another primary malignancy within 5 years prior to starting study treatment. Exceptions here are as follows: the disease under study; adequately treated basal or squamous cell carcinoma of the skin; cancer of the cervix in situ;
4. Active hepatitis B infection (If Hepatitis B surface antigen [HBsAg] or Hepatitis B core antibody [HBcAb] positive, then HBV-DNA must be < 20 IU/mL, and HBsAg-positive patients should have been treated with antiviral therapies as per the local guidelines);
5. Positive hepatitis C (HCV) RNA, Human Immunodeficiency Virus (HIV) antibody, Cytomegalovirus(CMV) DNA or syphilis serology;
6. Have received prior cell-based therapies such as targeted GPC3 therapy, TCR-T therapy, CAR-T therapy;
7. Inadequate bone marrow reserve or organ function;
8. History or current evidence of any condition or disease that could confound the results of the study or, in the opinion of Investigator, is not in the best interest of the patient to participate.
9. Pregnant or Breast-feeding women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of Ori-C101 | 1 year
  The MTD is defined as the highest dose with an observed incidence of DLT in no more than one out of six patients treated at a particular dose level.

SECONDARY OUTCOMES:
Objective Response Rate | 2 years
  Objective response is defined as the participants with a partial response (PR) or better by the RECIST1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Hunan Cancer Hospital, Changsha, Hunan
  - The first hospital of Jilin University, Changchun, Jilin
  - West China Hospital, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Lishui Central Hospital, Lishui, Zhejiang
  - Zhongshan Hospital Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No